CLINICAL TRIAL: NCT04450407
Title: A Phase 2, Randomized, Parallel, Open-Label Comparator-Controlled Trial to Evaluate the Safety and Efficacy of LY3209590 in Study Participants With Type 1 Diabetes Mellitus Previously Treated With Multiple Daily Injection Therapy
Brief Title: A Study of LY3209590 in Participants With Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17183; I8H-MC-BDCP (Other: Eli Lilly and Company); 2019-003589-41 (EudraCT Number)
Record Dates: First submitted 2020-06-26; First posted 2020-06-29 (Actual); Results first posted 2022-10-27 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-09

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — insulin degludec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LY3209590 Algorithm 1 (Paper) (Experimental): Algorithm 1 is a paper-based algorithm where dose adjustments were manually determined by the investigator based on fasting glucose and hypoglycemia data. LY3209590 was provided in a 20 milligram (mg) vial of reconstitutable lyophilized powder. Participants received individualized LY3209590 loading dose based on the basal insulin dose prior randomization and baseline fasting glucose by subcutaneous (SC) injection on day 1 followed by weekly adjustments for the first 12 weeks, then every 4 weeks, of a 26-week treatment period, to achieve target fasting glucose of <=100 milligrams per deciliter (mg/dL).
  Interventions: Drug: LY3209590
- LY3209590 Algorithm 2 (Digital) (Experimental): Algorithm 2 is a computer-based algorithm to determine dose adjustments. LY3209590 was provided in a 20 mg vial of reconstitutable lyophilized powder. Participants received individualized LY3209590 loading dose based on the basal insulin dose prior randomization and baseline fasting glucose by SC injection on day 1 followed by weekly adjustments for the first 12 weeks, then every 4 weeks, of a 26-week treatment period, to achieve target fasting glucose of <=100 mg/dL.
  As per protocol amendment (d) approved on 28-Oct-2020, this arm was terminated during the early enrollment phase due to technical issues with data entry.
  Interventions: Drug: LY3209590
- Insulin Degludec (Active Comparator): Insulin degludec was provided as 100 units/milliliter (U/mL) in a prefilled pen. Participants received individually adjusted doses once daily by SC injection with a starting dose same as basal insulin dose prior randomization, during the 26-week treatment period, to achieve target fasting blood glucose of <=100 mg/dL.
  Interventions: Drug: Insulin Degludec

INTERVENTIONS:
Drug: LY3209590 — Administered SC
  Arms: LY3209590 Algorithm 1 (Paper); LY3209590 Algorithm 2 (Digital)
Drug: Insulin Degludec — Administered SC
  Arms: Insulin Degludec

SUMMARY:
The reason for this study is to see if the study drug LY3209590 is safe and effective in participants with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a diagnosis of type 1 diabetes mellitus for at least 1 year
* Participants must have been using multiple daily injections without interruption for at least 3 months
* Participants must have HbA1c values of 5.6% to 9.5%, inclusive
* Participants must have a body mass index (BMI) of ≤35 kilograms per meter squared (kg/m²)

Exclusion Criteria:

* Have had more than 1 emergency room visit or hospitalization due to poor glucose control within 6 months prior to study screening
* Have any episodes of severe hypoglycemia and/or hypoglycemia unawareness within the 6 months prior to screening
* Have any of the following cardiovascular (CV) conditions: acute myocardial infarction, New York Heart Association Class III or IV heart failure, or cerebrovascular accident (stroke)
* Have acute or chronic hepatitis, or obvious clinical signs or symptoms of any other liver disease
* Have an estimated glomerular filtration rate (eGFR) <30 milliliters/minute/1.73 m²
* Have active or untreated cancer
* Are receiving chronic (>14 days) systemic glucocorticoid therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5hours, EST), Study Director — Eli Lilly and Company
Locations (54):
- United States (33):
  - John Muir Physician Network Clinical Research Center, Concord, California
  - Valley Endocrine, Fresno, Fresno, California
  - Coastal Metabolic Research Centre, Ventura, California
  - Barbara Davis Center for Childhood Diabetes, Aurora, Colorado
  - Denver Endocrinology, Diabetes & Thyroid Center, Englewood, Colorado
  - East Coast Institute for Research at The Jones Center, Jacksonville, Florida
  - Sun Coast Clinical Research, Inc, New Port Richey, Florida
  - Bayside Clinical Research, LLC, New Port Richey, Florida
  - Metabolic Research Institute, Inc., West Palm Beach, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - East Coast Institute for Research at The Jones Center, Macon, Georgia
  - Endocrine Research Solutions, Inc., Roswell, Georgia
  - Rocky Mountain Clinical Research, Idaho Falls, Idaho
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - Diabetes and Metabolism Associates, APMC, Metairie, Louisiana
  - Endocrine and Metabolic Consultants, Rockville, Maryland
  - Palm Research Center Tenaya, Las Vegas, Nevada
  - Southern Nh Diabetes and Endocrinology, Nashua, New Hampshire
  - Suny Health Science Center at Syracuse, Syracuse, New York
  - Lucas Research, Inc., Morehead City, North Carolina
  - PMG Research of Piedmont Healthcare, Statesville, North Carolina
  - PMG Research of Wilmington, Wilmington, North Carolina
  - Intend Research, LLC, Norman, Oklahoma
  - Holston Medical Group, Bristol, Tennessee
  - Univ Diab & Endo Consult, Chattanooga, Tennessee
  - Texas Diabetes & Endocrinology, P.A., Austin, Texas
  - Research Institute of Dallas, Dallas, Texas
  - Diabetes and Thyroid Center of Fort Worth, Fort Worth, Texas
  - Endocrine and Psychiatry Center, Houston, Texas
  - Southern Endocrinology Associates, Mesquite, Texas
  - Texas Diabetes & Endocrinology, P.A., Round Rock, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - Rainier Clinical Research Center, Renton, Washington
- Austria (3):
  - Universitätsklinikum Graz, Graz, Styria
  - Klinik Landstraße, Vienna
  - Zentrum für klinische Studien Dr Hanusch Gmbh, Vienna
- Germany (8):
  - Praxis Dr. Jörg Lüdemann, Falkensee, Brandenburg
  - InnoDiab Forschung Gmbh, Essen, North Rhine-Westphalia
  - Institut für Diabetesforschung GmbH Münster, Münster, North Rhine-Westphalia
  - Practice Dr.med. Denger and Dr.med. Pfitzner, Friedrichsthal, Saarland
  - Zentrum für klinische Studien, Saint Ingbert, Saarland
  - SMO.MD GmbH, Magdeburg, Saxony-Anhalt
  - RED-Institut GmbH, Oldenburg in Holstein, Schleswig-Holstein
  - Diabeteszentrum Hamburg West, Hamburg
- Puerto Rico (3):
  - Dr Altagracia Aurora Alcantara Gonzalez, Bayamón, PR
  - Advanced Clinical Research, LLC, Bayamón, PR
  - Martha Gomez Cuellar M.D., San Juan, PR
- Spain (7):
  - Hospital Universitario Virgen de la Victoria, Málaga, Andalusia
  - Hospital Quiron Infanta Luisa, Seville, Andalusia
  - Hospital Universitario de La Ribera, Alzira, Valencia
  - Complexo Hospitalario Universitario A Coruña, CHUAC, A Coruña
  - Centro Periférico de Especialidades Bola Azul, Almería
  - Clínica nuevas Tecnologías en Diabetes y Endocrinología, Seville
  - Hospital Universitario Virgen Macarena, Seville

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of LY3209590 in Participants With Type 1 Diabetes — https://trials.lillytrialguide.com/en-US/trial/5dp7c1Y8s5tS3GBCoGr1YO

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was initially designed as 3 arms: LY3209590 Algorithm 1 (Paper), LY3209590 Algorithm 2 (Digital), and Insulin Degludec. However, it was amended to terminate the "LY3209590 Algorithm 2 (Digital)" arm during early enrollment phase due to technical issues with data entry. Thus, this arm was excluded from the outcome measure analyses, but safety data was analysed and reported.
Groups:
- LY3209590 Algorithm 2 (Digital): Algorithm 2 is a computer-based algorithm to determine dose adjustments. LY3209590 was provided in a 20 mg vial of reconstitutable lyophilized powder. Participants received individualized LY3209590 loading dose based on the basal insulin dose prior randomization and baseline fasting glucose by SC injection on day 1 followed by weekly adjustments for the first 12 weeks, then every 4 weeks, of a 26-week treatment period, to achieve target fasting glucose of <=100 mg/dL.
Period: Overall Study
Arm/Group | LY3209590 Algorithm 1 (Paper) | LY3209590 Algorithm 2 (Digital) | Insulin Degludec
Started | 124 | 16 | 126
Received at Least One Dose of Study Drug | 123 | 16 | 126
Completed | 107 | 15 | 118
Not Completed | 17 | 1 | 8
Not completed — Withdrawal by Subject | 10 | 1 | 4
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Pregnancy | 1 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 0
Not completed — Investigational site terminated by sponsor | 3 | 0 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- LY3209590 Algorithm 1 (Paper): Algorithm 1 is a paper-based algorithm where dose adjustments were manually determined by the investigator based on fasting glucose and hypoglycemia data. LY3209590 was provided in a 20 mg vial of reconstitutable lyophilized powder. Participants received individualized LY3209590 loading dose based on the basal insulin dose prior randomization and baseline fasting glucose by SC injection on day 1 followed by weekly adjustments for the first 12 weeks, then every 4 weeks, of a 26-week treatment period, to achieve target fasting glucose of <=100 mg/dL.
- Insulin Degludec: Insulin degludec was provided as 100 U/mL in a prefilled pen. Participants received individually adjusted doses once daily by SC injection with a starting dose same as basal insulin dose prior randomization, during the 26-week treatment period, to achieve target fasting blood glucose of <=100 mg/dL.
- Total: Total of all reporting groups
Arm/Group | LY3209590 Algorithm 1 (Paper) | LY3209590 Algorithm 2 (Digital) | Insulin Degludec | Total
Number analyzed (Participants) | 124 | 16 | 126 | 266
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (14.8) | 53.4 (16.3) | 47.4 (13.7) | 46.4 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 4 | 48 | 102
  Male | 74 | 12 | 78 | 164
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 5 | 10 | 38
  Not Hispanic or Latino | 100 | 11 | 116 | 227
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 4 | 8
  White | 119 | 14 | 120 | 253
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Puerto Rico | 7 | 1 | 3 | 11
  Austria | 6 | 0 | 6 | 12
  United States | 80 | 15 | 84 | 179
  Germany | 16 | 0 | 18 | 34
  Spain | 15 | 0 | 15 | 30
Haemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: Percentage of HbA1c] — HbA1c is the glycosylated fraction of haemoglobin A. It is measured to identify average blood glucose concentration over prolonged periods of time. Population: All randomized participants with HbA1c data at baseline.
  Percentage of HbA1c
    number analyzed (Participants) | 124 | 16 | 125 | 265
    (all) | 7.52 (0.85) | 7.64 (0.70) | 7.45 (0.87) | 7.49 (0.85)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c)
Description: HbA1c is the glycosylated fraction of haemoglobin A. It is measured to identify average blood glucose concentration over prolonged periods of time. Least squares (LS) mean change from baseline was analysed by mixed model repeated measures (MMRM) model with treatment, country, visit, and treatment by visit interaction as fixed effects and the baseline HbA1c as a covariate.
Time Frame: Baseline, Week 26
Population: All participants randomized to either LY3209590 Algorithm 1 (Paper) or Insulin degludec, received at least one dose of study drug and had baseline, post-baseline HbA1c data prior to treatment discontinuation.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | LY3209590 Algorithm 1 (Paper) | Insulin Degludec
Number analyzed (Participants) | 118 | 123
Percentage of HbA1c | 0.04 (0.068) | -0.13 (0.065)
Statistical Analysis 1: Comparison: LY3209590 Algorithm 1 (Paper) vs Insulin Degludec; Test type: Non-Inferiority — The non-inferiority margin is 0.4%. Non-inferiority is achieved if the upper limit of the 90% CI (Confidence Interval) is below 0.4; LS Mean Difference = 0.17, 90% CI 2-sided [0.01 to 0.32]

2. Secondary Outcome: Change From Baseline in Fasting Serum Glucose
Description: LS mean change from baseline was analysed by mixed model repeated measures (MMRM) model with treatment, country, HbA1c stratum, visit, and treatment by visit interaction as fixed effects and the baseline fasting serum glucose as a covariate.
Time Frame: Baseline, Week 26
Population: All participants randomized to either LY3209590 Algorithm 1 (Paper) or Insulin degludec, received at least one dose of study drug and had baseline, post-baseline fasting serum glucose data prior to treatment discontinuation.
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | LY3209590 Algorithm 1 (Paper) | Insulin Degludec
Number analyzed (Participants) | 118 | 124
milligrams per deciliter (mg/dL) | -5.9 (5.65) | -16.7 (5.21)

3. Secondary Outcome: Change From Baseline in Bolus Insulin Dose
Description: Bolus insulin dose was the sum of doses for morning, midday, evening meals, snack and correction. LS mean change from baseline was analysed by MMRM model with treatment, country, HbA1c stratum, visit, and treatment by visit interaction as fixed effects and the baseline bolus insulin dose as a covariate.
Time Frame: Baseline, Week 26
Population: All participants randomized to either LY3209590 Algorithm 1 (Paper) or Insulin degludec, received at least one dose of study drug and had baseline, post-baseline bolus insulin dose data prior to treatment discontinuation.
Measure: Least Squares Mean (Standard Error); unit: Units per kilogram per day (U/kg/day)
Arm/Group | LY3209590 Algorithm 1 (Paper) | Insulin Degludec
Number analyzed (Participants) | 79 | 81
Units per kilogram per day (U/kg/day) | 0.04 (0.019) | 0.05 (0.018)

4. Secondary Outcome: Rate of Documented Hypoglycemia
Description: Documented hypoglycemia is defined as any time a participant reports a self-monitoring blood glucose <54 mg/dL (3.0 millimole per liter (mmol/L)). Negative binomial model using baseline hypoglycaemia incidence, baseline HbA1c and treatment as independent variables was performed to estimate the event rate. Data presented is group mean. Group Mean is estimated by first taking the inverse link function on individual participant covariates, then averaging over all participants.
Time Frame: Baseline through Week 26
Population: All participants randomized to either LY3209590 Algorithm 1 (Paper) or Insulin degludec, received at least one dose of study drug.
Measure: Mean (Standard Error); unit: Events per participant per year
Arm/Group | LY3209590 Algorithm 1 (Paper) | Insulin Degludec
Number analyzed (Participants) | 123 | 126
Events per participant per year | 20.7 (2.27) | 18.4 (2.00)

5. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Time Curve (AUC) of LY3209590
Description: AUC of LY3209590 was calculated for individual participants using the participant's Week 26 LY3209590 dose amount and the estimated clearance value.
Time Frame: Week 26
Population: All participants randomized to LY3209590 Algorithm 1 (Paper), received at least one dose of study drug and had evaluable PK data at Week 26.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomole*hour per Liter (nmol*hr/L)
Arm/Group | LY3209590 Algorithm 1 (Paper)
Number analyzed (Participants) | 99
Nanomole*hour per Liter (nmol*hr/L) | 3520 (53)

ADVERSE EVENTS:
Time Frame: Baseline to Follow-up (up to 31 weeks)
Description: All randomized participants. Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
Arm/Group | LY3209590 Algorithm 1 (Paper) | LY3209590 Algorithm 2 (Digital) | Insulin Degludec
All-Cause Mortality (participants affected / at risk) | 0/124 | 0/16 | 0/126
Serious Adverse Events (participants affected / at risk) | 5/124 | 0/16 | 4/126
Other Adverse Events (participants affected / at risk) | 21/124 | 7/16 | 11/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LY3209590 Algorithm 1 (Paper) (N=124) | LY3209590 Algorithm 2 (Digital) (N=16) | Insulin Degludec (N=126)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Maternal exposure during pregnancy (Injury, poisoning and procedural complications) | 1/50 (1) | 0/4 (0) | 0/48 (0)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (2)
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY3209590 Algorithm 1 (Paper) (N=124) | LY3209590 Algorithm 2 (Digital) (N=16) | Insulin Degludec (N=126)
Injection site bruising (General disorders) | 1 (1) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 2 (2) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 3 (4) | 1 (1) | 1 (1)
Onychomycosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (2) | 1 (1)
Sars-cov-2 test positive (Investigations) | 2 (2) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 10 (14) | 0 (0) | 5 (5)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 4 (4) | 1 (1) | 3 (3)

LIMITATIONS AND CAVEATS:
The study was initially designed as 3 arms: LY3209590 Algorithm 1 (Paper), LY3209590 Algorithm 2 (Digital), and Insulin Degludec. However, it was amended to terminate the "LY3209590 Algorithm 2 (Digital)" arm during early enrollment phase due to technical issues with data entry. Thus, this arm was excluded from the outcome measure analyses, but safety data was analysed and reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-10-28): https://cdn.clinicaltrials.gov/large-docs/07/NCT04450407/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-08): https://cdn.clinicaltrials.gov/large-docs/07/NCT04450407/SAP_001.pdf